CLINICAL TRIAL: NCT02117557
Title: A Prospective Randomized Controlled Trial Comparing Transumbilical Single Incision Versus Conventional Laparoscopic Surgery for Colorectal Cancer
Brief Title: Safety Study of Transumbilical Single Incision Versus Conventional Laparoscopic Surgery for Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guoxin Li (Other)
Responsible Party: Sponsor-Investigator, Guoxin Li, M.D., Ph.D., Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NFGS-SILS-01
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Colorectal Cancer
Keywords: Single-incision; Laparoscopy; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single incision laparoscopic surgery (Experimental): Transumbilical single incision laparoscopic surgery will be performed for patients in this group.And addition of only one trocar through the stoma for drainage tube is allowed.
  Interventions: Procedure: Single incision laparoscopic surgery
- Conventional laparoscopic surgery (Active Comparator): Conventional laparoscopic surgery for colorectal cancer will be performed for patients in this group.
  Interventions: Procedure: Conventional laparoscopic surgery

INTERVENTIONS:
Procedure: Single incision laparoscopic surgery
  Other Names: SILS
  Arms: Single incision laparoscopic surgery
Procedure: Conventional laparoscopic surgery
  Other Names: CLS
  Arms: Conventional laparoscopic surgery

SUMMARY:
* Compared with traditional open colectomy, laparoscopic surgery is associated with less pain, earlier recovery, and better cosmetic outcome, and its short- and long-term oncologic outcomes have been demonstrated.
* In experienced surgeons' hands, single incision laparoscopic surgery is increasingly performed for colorectal disease, and even for malignant lesion because of its reduced incision-associated morbidity and scarring.
* However, the safety and efficacy of single incision laparoscopic surgery for colorectal cancer has not yet been evaluated. Thus, the prospective randomized trial comparing single incision versus conventional laparoscopic surgery for colorectal cancer is needed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years < age < 80 years
* Tumor located in rectosigmoid (defined as 10- to 30-cm from the anal verge)
* Pathological rectosigmoid carcinoma
* Preoperative T stage ranging from T1 to T4a according to the 7th Edition of AJCC Cancer Staging Manual
* Tumor size of 5 cm or less; 6) ECOG score is 0-1
* ASA socre is Ⅰ-Ⅲ
* Informed consent

Exclusion Criteria:

* Body mass index (BMI) >30 kg/m2
* Pregnant woman or lactating woman
* Severe mental disease
* Previous abdominal surgery
* Emergency operation due to complication (bleeding, perforation or obstruction) caused by colorectal cancer
* Requirement of simultaneous surgery for other disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Early morbidity rate | 30 days
  The early morbidity rate is defined as the event observed during operation and within 30 days after surgery,

SECONDARY OUTCOMES:
Operative outcomes | intraoperative
  Operative time, estimated blood loss and incision length are recorded.
Pathological outecomes | 5 days
  Tumor size, length of proximal and distal margin and lymph nodes harvested are used to assess oncological resection.
Postoperative recovery course | 14 days
  Time to first ambulation, flatus, liquid diet, soft diet, and duration of hospital stay are used to assess the postoperative recoverty course.
Pain score | 14 days
  Postoperative pain is recorded using the visual analog scale (VAS) pain score tool on postoperative day 1, 2, 3 and the day of discharge.
Cosmetic assessment | 14 days
  Cosmetic assessment is perform using body image scale and cosmetic scale.
3-year disease free survival rate | 36 months
5-year overall survival rate | 60 months
Inflammatory and immune response | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Guoxin Li, M.D., PH.D., Principal Investigator — Nanfang Hospital, Southern Medical University, China
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bucher P, Pugin F, Morel P. Single-port access laparoscopic radical left colectomy in humans. Dis Colon Rectum. 2009 Oct;52(10):1797-801. doi: 10.1007/DCR.0b013e3181b551ce. PMID 19966617
- [Background] Gash KJ, Goede AC, Chambers W, Greenslade GL, Dixon AR. Laparoendoscopic single-site surgery is feasible in complex colorectal resections and could enable day case colectomy. Surg Endosc. 2011 Mar;25(3):835-40. doi: 10.1007/s00464-010-1275-8. Epub 2010 Aug 24. PMID 20734083
- [Background] Lim SW, Kim HJ, Kim CH, Huh JW, Kim YJ, Kim HR. Umbilical incision laparoscopic colectomy with one additional port for colorectal cancer. Tech Coloproctol. 2013 Apr;17(2):193-9. doi: 10.1007/s10151-012-0900-z. Epub 2012 Sep 19. PMID 22991135
- [Background] Hirano Y, Hattori M, Douden K, Shimizu S, Sato Y, Maeda K, Hashizume Y. Single-incision plus one port laparoscopic anterior resection for rectal cancer as a reduced port surgery. Scand J Surg. 2012;101(4):283-6. doi: 10.1177/145749691210100411. PMID 23238505
- [Derived] Zhang X, Yuan H, Tan Z, Li G, Xu Z, Zhou J, Fu J, Wu M, Xi J, Wang Y. Long-term outcomes of single-incision plus one-port laparoscopic surgery versus conventional laparoscopic surgery for rectosigmoid cancer: a randomized controlled trial. BMC Cancer. 2023 Dec 7;23(1):1204. doi: 10.1186/s12885-023-11500-2. PMID 38062421
- [Derived] Wang Y, Deng H, Mou T, Li J, Liu H, Zhou H, Li G. Short-term outcomes of single-incision plus one-port laparoscopic versus conventional laparoscopic surgery for rectosigmoid cancer: a randomized controlled trial. Surg Endosc. 2019 Mar;33(3):840-848. doi: 10.1007/s00464-018-6350-6. Epub 2018 Jul 13. PMID 30006846
- [Derived] Wang Y, Liu R, Zhang Z, Xue Q, Yan J, Yu J, Liu H, Zhao L, Mou T, Deng H, Li G. A safety study of transumbilical single incision versus conventional laparoscopic surgery for colorectal cancer: study protocol for a randomized controlled trial. Trials. 2015 Nov 30;16:539. doi: 10.1186/s13063-015-1067-5. PMID 26620555